CLINICAL TRIAL: NCT02384694
Title: ZumBeat: Effekte Eines Rhythmusorientierten Aeroben Tanz-Bewegungsprogrammes für Postmenopausale Frauen Mit Metabolischem Syndrom
Brief Title: Effects of a Zumba Dance Program for Postmenopausal Women With Metabolic Syndrome
Acronym: ZumBeat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Prof. Arno Schmidt-Trucksäss, MD, MA, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2014-033
Record Dates: First submitted 2015-02-27; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Metabolic Syndrome
Keywords: cardiorespiratory fitness; weight; quality of life; depression; menopausal symptoms; exercise barriers; executive functions
MeSH Terms: conditions — Metabolic Syndrome; Body Weight; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Zumba dance intervention
  Interventions: Other: Zumba dance

INTERVENTIONS:
Other: Zumba dance — Twelve weeks, 3 times weekly 1 hour training

SUMMARY:
The aim of this study is to examine the effects of a 12-week Zumba dance intervention on fitness, anthropometric and psychometric parameters and eating behavior.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (Age 45-65)
* waist of >94 cm or BMI > 30kg/m2
* not physically active >1x/week for 20 minutes
* written consent before the start of the study

Exclusion Criteria:

* involvement in other clinical studies
* unable to participate at the dance lessons
* medical contraindications for the intervention or increased risk for exercise participation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
VO2peak (=peak oxygen consumption) | VO2peak will be assessed at T1 and T12 (baseline and after 12 weeks of intervention)
  The VO2peak will be assessed for every participant during a treadmill spirometry at baseline and follow-up using a mask and calibrated gas measuring devices applying a standardized protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof. Dr., Principal Investigator — Sports and Exercise Medicine, Department of Sports, Exercise and Health, University of Basel
Locations (1):
- Department for Sports, Exercise and Health, Sports and Exercise Medicine, University of Basel, Basel, Switzerland